CLINICAL TRIAL: NCT06330467
Title: Prevalence of Dissociative Identity Disorder in At-risk Outpatient Groups Reporting Childhood Trauma.
Acronym: IDENTITY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Psychothérapique de Nancy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A02442-43; RIPH 2023-02 (Registry Identifier: sponsor's internal reference)
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Dissociative Disorder
Keywords: Dissociative Identity Disorder (DID); Psychosis; Functional Dissociative Crises (FDC); Complex PTSD; Borderline
MeSH Terms: conditions — Dissociative Disorders; Dissociative Identity Disorder; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: 3 groups : borderline, early psychosis and FDC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Borderline (Other): Borderline patients
  Interventions: Diagnostic Test: psychometric assessment; Diagnostic Test: semi-structured clinical interview
- Functional Dissociative Crises (FDC) (Other): FDC patients
  Interventions: Diagnostic Test: psychometric assessment; Diagnostic Test: semi-structured clinical interview
- Early psychosis (Other): Early psychosis patients : mental state at risk for psychosis and first psychotic episode
  Interventions: Diagnostic Test: psychometric assessment; Diagnostic Test: semi-structured clinical interview

INTERVENTIONS:
Diagnostic Test: psychometric assessment — Psychometric testing to assess trauma and dissociative disorders, and in particular dissociative identity disorder.
Diagnostic Test: semi-structured clinical interview — Semi-structured interview for the assessment of dissociative disorders (SCID-D : Semi-structured Clinical Interview for diagnosing DSM-5 and ICD-11 Dissociative Disorders)

SUMMARY:
The investigators will study the prevalence of dissociative identity disorder (DID) in three populations at risk in cases of childhood psychotrauma : patients with a diagnosis of borderline personality, patients with a diagnosis of functional dissociative crises (FDC) and patients with early psychosis.

The investigators will also study the prevalence of other dissociative disorders and the frequency of complex post-traumatic stress disorder.

The investigators will also look for correlations between the type of maltreatment in childhood, the age of onset of trauma and the type of diagnosis of dissociative disorders.

The investigators hope to include 150 borderline patients, 150 FDC patients and 50 early psychosis patients.

Data collection will be done via a psychometric administration of 7 self-completion questionnaires as well as the completion of the SCID-D semi-structured interview.

ELIGIBILITY:
I - Inclusion Criteria:

I-1: For all groups:

* Male or female
* Age > or = 18
* Enrolled in or benefiting from a social security scheme
* Patient fluent in French
* Patient willing to undergo a psychological evaluation between 1h30 and 3h30
* Patient with a known history of psychotrauma in childhood before the age of 18 (sexual abuse, mistreatment, school harassment, natural disasters, attacks, etc.).
* Patient having received and understood complete information on the organization of the research and having given written free and informed consent prior to participation in the study.

I-2 : Patients in the borderline group

* Patients with main diagnosis of emotionally labile personality
* Patients with at least one psychiatric hospitalization in the last 3 years

I-3 : Patients in the early psychosis group

Patient with a diagnosis of mental state at risk of psychosis according to the criteria defined by CAARMS (Comprehensive Assessment of At Risk Mental State) OR Patients diagnosed with a first psychotic episode on an outpatient basis or following a hospital stay

I-4 : Patients in the functional dissociative crises group

Patients diagnosed with functional dissociative crises by a specialized epileptologist

II- Non-inclusion criteria

* Impairment of the subject making it difficult or not impossible to participate in the trial or to understand the information provided to him/her
* Patients with specific difficulties in understanding SCID-D questions
* Psychiatric condition requiring hospitalization
* Patients with symptoms of recent toxic consumption (alcohol, cannabis, other ...) disrupting assessment responses
* Patient taking part in a pharmacological study involving a pro-dissociative molecule of the psychedelic type
* Pregnant, parturient or nursing mothers
* Person deprived of liberty by judicial or administrative decision
* Person in a life-threatening emergency
* An adult under legal protection (guardianship, curatorship, safeguard of justice)
* Person unable to give consent and not subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-08-18 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
SCID-D : Semi-structured Clinical Interview for diagnosing DSM-5 and ICD-11 Dissociative Disorders / DSM = Diagnostic and Statistical Manual of Mental Disorders / ICD = International Classification of Diseases | Inclusion visit
  assesses the dissociative identity disorder

SECONDARY OUTCOMES:
SCID-D : Semi-structured Clinical Interview for diagnosing DSM-5 and ICD-11 Dissociative Disorders | Inclusion visit
  assesses the 4 others domains of dissociative disorders
CTQ-28 : Childhood Trauma Questionnaire | Inclusion visit
  assesses history of childhood abuse and childhood trauma. For the CTQ-28, the overall score is not really relevant, but rather the scores for each type of abuse. For each type of maltreatment, there are differences in severity, ranging from "none" to "severe", with threshold scores for each level. In fact, there is no real overall minimum or maximum score.
life events inventory DSM-5 | Inclusion visit
  assesses history of potentially traumatic life events. There is no numerical score, it's simply an inventory of potentially traumatic life events.
PCL-5 : Posttraumatic stress disorder CheckList-5 | Inclusion visit
  assess the Post Traumatic Stress Disorder. For the PCL-5, the threshold score is 33, so a score of 33 or more suggests the presence of PTSD : the higher the score, the greater the symptomatology. The score is not a value used for interpretation purposes. The investigators use only threshold scores, or diagnostic criteria.
ITQ : International Trauma Questionnaire | Inclusion visit
  assesses simple and complex post-traumatic stress syndrome. For the ITQ, there is no real numerical score; the diagnosis of PTSD or complex PTSD is made on the basis of the diagnostic criteria met.
  Scores are not given with numbers, but only with the presence or absence of simple or complex PTSD. There is no minimum or maximum score.
SDQ-20 : Somatoform Dissociative questionnaire | Inclusion visit
  assess somatoform dissociation. For the SDQ-20, the threshold score is 28, and there are no levels of severity: the higher the score, the more severe the somatoform dissociative disorders. However, the score should be treated with caution, as if the symptoms reported by the patient are explained by a medical cause, we cannot conclude that dissociative disorders are present despite the score.
DIS-Q : Dissociation Questionnaire | Inclusion visit
  assess the dissociative disorders. For the DIS-Q, the threshold score is 2.5. The score is not a value used for interpretation purposes. The investigators use only threshold scores, or diagnostic criteria.
DES : Dissociative Experience Scale | Inclusion visit
  assess the dissociative disorder. For the DES, there is a threshold score of 15, and the higher the score, the more severe the dissociative disorders, but there are no multiple levels of severity. The score is not a value used for interpretation purposes. The investigators use only threshold scores, or diagnostic criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Coraline HINGRAY, Principal Investigator — Centre Psychothérapique de Nancy
Locations (3):
- France (3):
  - Centre Psychothérapique de Nancy - CLIP, Nancy
  - Centre Psychothérapique de Nancy - CMP Jacquard et Des Près, Nancy
  - CHRU Nancy - Neurology department, Nancy

IPD SHARING:
Plan to Share IPD: No